CLINICAL TRIAL: NCT04216888
Title: Biomarkers of Response to Ketamine in Depression
Brief Title: Biomarkers of Response to Ketamine in Depression: MRI and Blood Assays Before and After Open Label Intranasal Ketamine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dan Iosifescu (Other)
Responsible Party: Sponsor-Investigator, Dan Iosifescu, Director of Clinical Reserach, Nathan Kline Institute for Psychiatric Research
Organization: Nathan Kline Institute for Psychiatric Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KetBiomarkers
Record Dates: First submitted 2019-08-26; First posted 2020-01-03 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental): Open label intranasal ketamine
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Intranasal administration of 40mg ketamine hydrochloride using an intranasal mucosal atomization device

SUMMARY:
This pilot study aims to identify predictors of response to intranasal ketamine treatment in patients with treatment-resistant depression. Participants will give a sample of blood and undergo magnetic resonance imaging before and after a single intranasal ketamine treatment. Participants will subsequently receive a second intranasal ketamine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years of age, inclusive, at screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Ability to participate in MRI (no history of claustrophobia, no presence of metallic foreign bodies incompatible with MRI, as assessed with MRI checklist and clinical interview).
4. Diagnosed with Major Depressive Disorders (MDD), single or recurrent, and currently experiencing a major depressive episode (MDE) of at least eight weeks in duration, prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). The diagnosis of MDD will be made by a site psychiatrist and supported by the Structured Clinical Interview for DSM-5 (SCID-5).
5. Has a history of treatment-resistant depression (TRD), as assessed by the investigator using the Mass General Hospital Antidepressant Treatment History Questionnaire (MGH ATRQ). TRD is defined as failure to achieve a satisfactory response (e.g., less than 50% improvement of depression symptoms), as perceived by the participant, to at least 1 "treatment course" of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration (including the current antidepressant treatment). The adequacy of dose and duration of the antidepressant therapy will be determined as per the MGH ATRQ criteria.
6. Depression is of at least "moderate" severity, as determined by a Clinical Global Impression-Severity scale (CGI-S) score greater than or equal to 4).
7. In good general health, as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and electrocardiogram (ECG).
8. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   a. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or b. Childbearing potential, and meets the following criteria: i. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.

   ii. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at baseline, prior to receiving ketamine treatment.

   iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
9. Body mass index between 18-35 kg/m2.
10. Concurrent benzodiazepine therapy will be allowed if the dose is less than or equal to 2mg of lorazepam (or the equivalent) per day and stable for the past 4 weeks.

Exclusion Criteria:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. Current diagnosis of a substance use disorder, except for nicotine dependence, at screening or within 6 months prior to screening.
5. History of bipolar disorder, schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
6. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within 5 years of screening.
7. In the judgment of the investigator, the subject is considered at significant risk for suicidal behavior during his/her participation in the study.
8. Has dementia, delirium, amnestic, or any other cognitive disorder.
9. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to the study clinician.
10. Current episode of:

    1. Hypertension, Stage 1 as defined by a systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening (Visit 1) or within 1.5 hours prior to ketamine administration on two of three measurements (standing and supine) at least 15 minutes apart.
    2. Recent myocardial infarction (within one year) or a history of myocardial infarction.
    3. Syncopal event within the past year.
    4. Congestive heart failure (CHF): New York Heart Association Criteria >Stage 2
    5. Angina pectoris.
    6. Heart rate <45 or >110 beats per minute at screening or Visit 3 ( first ketamine administration).
    7. QTcF (Fridericia-corrected) ≥450 msec at screening or Visit 3 (first ketamine administration).
11. Chronic lung disease excluding asthma.
12. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention which, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS, or history of significant head trauma within the past 2 years.
13. Presents with any of the following lab abnormalities:

    1. Thyroid stimulating hormone (TSH) outside of the normal limits and clinically significant as determined by the investigator. Free thyroxine (T4) levels may be measured if TSH level is high. Subject will be excluded if T4 level is clinically significant.
    2. Patients with diabetes mellitus fulfilling any of the following criteria:

    i. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening.

    ii. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.

    iii. Not under physician care for diabetes mellitus. iv. Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.

    c. Any other abnormal laboratory result(s), clinically significant in the opinion of the investigator, at the time of the screening.
14. History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than 2 months prior to screening. (Subjects on a stable dosage of thyroid replacement medication for at least 2 months or more prior to screening are eligible for enrollment.)
15. History of hyperthyroidism which was treated (medically or surgically) less than 6 months prior to screening.
16. History of positive screening urine test for drugs of abuse at screening: cannabinoids (if the patient has a legitimate medical prescription for cannabis, patient must agree to abstain during the entirety of the study and to have a negative test at baseline), cocaine, amphetamines, barbiturates, opiates (unless use is in accordance with guidance provided in Appendix 1, table of allowed and excluded medications).
17. Patients with exclusionary laboratory values (see Table 1) or requiring treatment with exclusionary concomitant medications (see Appendix 1).
18. Patients with a history of narrow angle glaucoma.
19. Liver or renal Function Tests (LFTs) which meet the exclusion criteria in Table 1, or a history of hepatic or renal dysfunction.
20. Self-reported history of a ketamine or hallucinogen abuse or misuse.

TABLE 1: EXCLUSIONARY SAFETY VALUES OF POTENTIAL CLINICAL CONCERN Hematology Leukocytes <2 or >17.5 x 103/mm3 Platelets <75 or >700 x 103/mm3 Chemistry Total bilirubin >2 times the upper limit of the reference range AST* >2.5 times upper limit of the reference range ALT* >2.5 times upper limit of the reference range GGT* >2.5 times upper limit of the reference range Alk Phosphatase* >2.5 times upper limit of the reference range Creatinine >1.3 times upper limit of the reference range BUN/Urea >1.3 times upper limit of the reference range Glucose < 70 mg/dl or >2 times the limits of the reference range Uric acid >1.5 times upper limit of the reference range

*LFTs higher than 2.5 times ULN will be exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery and Asberg Depression Rating Scale (MADRS) | 24 hours
  Montgomery and Asberg Depression Rating Scale (MADRS), with scores ranging from 0-60; higher scores indicate more severe depression. Change will be calculated as the difference between MADRS scores at baseline (day of but prior to first ketamine treatment) and a 24 hour follow-up visit.
Cortical thickness | within 48 hours (pretreatment)
  We will test for baseline differences in cortical thickness which differentiate responders and non-responders to ketamine.

SECONDARY OUTCOMES:
Neural response to affective stimuli | within 48 hours (post treatment)
  We will test for baseline differences in functional anisotropy of white matter tracts which differentiate responders and non-responders to ketamine.
Neural response to affective stimuli | within 48 hours (pretreatment)
  We will test for changes in cognitive control network (CCN) activation and functional connectivity (FC) of anterior aspects of the CCN (middle frontal gyrus [MFG] and dorsal anterior cingulate cortex [dACC]) during an emotional regulation task.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, MSc, Principal Investigator — Nathan Kline Institute
Locations (1):
- Nathan Kline Institute, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: No